CLINICAL TRIAL: NCT03272269
Title: A Phase I Placebo-controlled, Double-blind, Dose Escalation Clinical Trial to Evaluate the Safety and Immune Responses of Imcyse's IMCY-0098 in Patients With Recent Onset Type 1 Diabetes
Brief Title: Study of IMCY-0098 in Patients With Recent Onset Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imcyse SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IMCY-T1D-001
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus type 1; Autoimmune disease; Immunotherapy; Diabetes treatment; Residual beta cell function; Adult patients
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1, low dose (Experimental): 4 SC injections of IMCY-0098 or Placebo
  Interventions: Drug: IMCY-0098; Other: Placebo
- Cohort 2, medium dose (Experimental): 4 SC injections of IMCY-0098 or Placebo
  Interventions: Drug: IMCY-0098; Other: Placebo
- Cohort 3, high dose (Experimental): 4 SC injections of IMCY-0098 or Placebo
  Interventions: Drug: IMCY-0098; Other: Placebo

INTERVENTIONS:
Drug: IMCY-0098 — Small synthetic peptide for SC admin. Solvent: alum hydroxide
  Other Names: Imotope
Other: Placebo — Solvent: alum hydroxide

SUMMARY:
This clinical study will evaluate the safety of an innovative approach expected to be disease-modifying by stopping the auto-immune-mediated destruction of islet β-cells in the pancreas. Three doses of the investigational product will be tested in successive cohorts. Although safety is the first objective of this study, we will gather efficacy data and perform a set of immunological tests to further understand the mechanism of action of this new approach in young adults with recent onset type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 30 years of age
2. Initial diagnosis of Type 1 diabetes according to ADA/WHO criteria within the past 6 months
3. Insulin requirement, as determined by the investigator
4. Presence of at least one autoantibody (GAD65, IA-2, or ZnT8)
5. Fasting C-peptide at screening >0.2 nmol/L and/or stimulated C-peptide ≥ 0,4 nmol/L.
6. HLADR3-positive and/or HLADR4-positive
7. Willingness to undergo the insulin treatment prescribed by the physician
8. Body mass index (BMI) between 17-28 kg/m2 at screening
9. Fully informed written consent obtained
10. Males with reproductive potential should use barrier method of contraception (condom) from screening up to 90 days after last treatment with investigational product.
11. Women of childbearing potential should use an highly effective contraception method from screening and for the whole duration of the study.

Exclusion Criteria:

1. Ongoing or planned pregnancy during the whole duration of the study or lactation
2. Presence of significant medical conditions in particular chronic liver condition, chronic hematological disease, renal dysfunction of grade 2 or more according to the World Health Organization (WHO) Toxicity Scale .
3. Has any current signs or symptoms of infection at entry or within 2 weeks of entry or has received intravenous antibiotics within 2 months prior to the first planned administration of the study product
4. Has received any live, attenuated vaccine within 3 months prior to the first planned administration of the study product (i.e. oral poliomyelitis vaccine, measles-mumps-rubella vaccine, yellow fever vaccine, Japanese encephalitis vaccine, dengue vaccine, rotavirus vaccine, varicella vaccine, live-attenuated zoster vaccine, Bacillus Calmette-Guérin [BCG] vaccine, oral typhoid vaccine)
5. History of, or current malignancy (except excised basal cell skin cancer)
6. Clinical evidence of a diabetes-related complication that could interfere with patient's participation/completion of study
7. Primary or secondary immune deficiency disorders
8. Human Immunodeficiency virus (HIV), chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
9. Presence at screening of abnormal laboratory values grade 2 or more according to the World Health Organization (WHO) Toxicity Scale
10. Anti-diabetic treatments other than insulin in the week prior to first study drug administration
11. Ongoing treatment with immunosuppressive agents or treatment within the past year with the exception of topical or intra nasal corticosteroids.
12. Treatment with immunotherapy within the past 3 months
13. Treatment with an investigational drug within the past 3 months
14. Patients with a known hypersensitivity to any component of the drug product should be excluded from the study
15. Patients under treatment with statins at the time of screening.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of all adverse events reported for subjects | up to 24 weeks
  Safety assessed through measurement and comparison of any reactions or hypersensitivity to IMCY-0098 injection vs placebo. Number of adverse events will also be compared between groups with the addition of safety monitoring blood tests

SECONDARY OUTCOMES:
Assessment of residual beta cell function and markers of metabolic control | up to 24 weeks
  Measured by a change in stimulated C-peptide production, daily insulin usage, glycated haemoglobin levels and glucose levels and excursions from baseline and between groups

OTHER OUTCOMES:
Assessment of T lymphocyte immune response to IMCY-0098 | up to 24 weeks
  Comparison of changes in IMCY-0098 specific T lymphocyte responses longitudinally following peptide treatment and versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vandepapelière, MD, Study Director — Imcyse SA; Christian Boitard, MD, Principal Investigator — Hôpital Cochin, Paris, France
Locations (17):
- Belgium (3):
  - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
- Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark
- CHU de Nantes, Hôpital Laennec, Nantes, France
- GWT-TUD GmbH, Dresden, Germany
- Lithuania (2):
  - Klaipeda University Hospital, Klaipėda
  - University Hospital Santaros Klinikos, Vilnius
- Sweden (2):
  - Clinical Trial Center, CTC, Gothenburg
  - ProbarE Stockholm, Stockholm
- United Kingdom (7):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff University, Cardiff
  - Royal Devon and Exeter NHS Trust, Exeter
  - Guy's and St. Thomas NHS Trust, London
  - St. Bartholomew's Hospital (Barts Health NHS Trust), London
  - Newcastle University, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlier VA, VanderElst L, Janssens W, Jacquemin MG, Saint-Remy JM. Increased synapse formation obtained by T cell epitopes containing a CxxC motif in flanking residues convert CD4+ T cells into cytolytic effectors. PLoS One. 2012;7(10):e45366. doi: 10.1371/journal.pone.0045366. Epub 2012 Oct 9. PMID 23056200
- [Background] Malek Abrahimians E, Carlier VA, Vander Elst L, Saint-Remy JM. MHC Class II-Restricted Epitopes Containing an Oxidoreductase Activity Prompt CD4(+) T Cells with Apoptosis-Inducing Properties. Front Immunol. 2015 Sep 2;6:449. doi: 10.3389/fimmu.2015.00449. eCollection 2015. PMID 26388872
- [Background] Malek Abrahimians E, Vander Elst L, Carlier VA, Saint-Remy JM. Thioreductase-Containing Epitopes Inhibit the Development of Type 1 Diabetes in the NOD Mouse Model. Front Immunol. 2016 Mar 2;7:67. doi: 10.3389/fimmu.2016.00067. eCollection 2016. PMID 26973647
- [Derived] Van Rampelbergh J, Achenbach P, Leslie RD, Kindermans M, Parmentier F, Carlier V, Bovy N, Vanderelst L, Van Mechelen M, Vandepapeliere P, Boitard C. First-in-human, double-blind, randomized phase 1b study of peptide immunotherapy IMCY-0098 in new-onset type 1 diabetes: an exploratory analysis of immune biomarkers. BMC Med. 2024 Jun 21;22(1):259. doi: 10.1186/s12916-024-03476-y. PMID 38902652
- [Derived] Van Rampelbergh J, Achenbach P, Leslie RD, Ali MA, Dayan C, Keymeulen B, Owen KR, Kindermans M, Parmentier F, Carlier V, Ahangarani RR, Gebruers E, Bovy N, Vanderelst L, Van Mechelen M, Vandepapeliere P, Boitard C. First-in-human, double-blind, randomized phase 1b study of peptide immunotherapy IMCY-0098 in new-onset type 1 diabetes. BMC Med. 2023 May 24;21(1):190. doi: 10.1186/s12916-023-02900-z. PMID 37226224
- See also: Registre belge du diabète — http://www.bdronline.be/index.php?n=169&id=267&sid=267&taal=F&mnav=2
- See also: Belgisch diabetes register — http://www.bdronline.be/index.php?n=164&id=265&sid=265&taal=N&mnav=2
- See also: Research study for people with Type 1 Diabetes: EXALT — http://www.address2.org/t1d-studies/